CLINICAL TRIAL: NCT05036980
Title: Randomized, Double-Blind, Placebo-Controlled, Crossover Study of Trans Sodium Crocetinate in Healthy Volunteers Exercising at Altitude
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200-302
Record Dates: First submitted 2021-07-30; First posted 2021-09-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers With Induced Hypoxia
MeSH Terms: interventions — trans-sodium crocetinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5 mg/kg Trans Sodium Crocetinate (Experimental): Subjects will receive a single IV bolus dose of 0.5 mg/kg TSC. Subjects will also receive a single IV dose of normal saline as placebo, thereby serving as their own control.
  Interventions: Drug: Trans Sodium Crocetinate
- 1.5 mg/kg Trans Sodium Crocetinate (Experimental): Subjects will receive a single IV bolus dose of 1.5 mg/kg TSC. Subjects will also receive a single IV dose of normal saline as placebo, thereby serving as their own control.
  Interventions: Drug: Trans Sodium Crocetinate
- 2.5 mg/kg Trans Sodium Crocetinate (Experimental): Subjects will receive a single IV bolus dose of 2.5 mg/kg TSC. Subjects will also receive a single IV dose of normal saline as placebo, thereby serving as their own control.
  Interventions: Drug: Trans Sodium Crocetinate

INTERVENTIONS:
Drug: Trans Sodium Crocetinate — Single IV bolus

SUMMARY:
This is a randomized, placebo-controlled, crossover study of Trans Sodium Crocetinate (TSC) in healthy volunteers, age 18-40 (inclusive), exercising at altitude. The primary objective is to determine the effect of (TSC) on partial pressure of oxygen (PaO2) and maximal oxygen consumption (VO2 max); the secondary objective is to assess the effect of TSC on oxygen saturation (SpO2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females ages 18-40
2. Non-smoking
3. Able to provide informed consent and agree to adhere to all study visits and requirements.
4. Females of childbearing potential must have a negative blood pregnancy test at screening and agree to use one of the accepted contraceptive regimens, or a double method of birth control during the study and at least 30 days after the last dose of study drug.
5. Males who engage in sexual activity that has the risk of pregnancy must agree to use a double barrier method and agree not to donate sperm during the study and for at least 90 days after the last dose of study drug

Exclusion Criteria:

1. Allergy to study medication
2. Pregnant or breast feeding
3. Received investigational medicine (IMP) within past 30 days
4. VO2 max < 35 mL/kg/min (male), < 30 mL/kg/min (female) at screening
5. Abnormal pulmonary function testing at screening
6. Surgery or hospitalization in past 3 months determined by the PI to be clinically relevant
7. History of ongoing alcohol or substance abuse
8. Known cardiovascular disease, including treated or untreated hypertension
9. Respiratory disease and/or any other significant medical condition, including psychiatric disorders
10. Clinically significant abnormality on ECG per PI discretion
11. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening
12. Plasma donation within 7 days prior to screening
13. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening
14. History of smoking
15. Urine screen positive for drugs or positive breathalyzer for alcohol (at screening and Treatment Visit Day 1)
16. History of seizures
17. Previous pneumothorax or pneumomediastinum
18. Hypo/Hyperglycemia
19. Diabetes
20. Regularly taking medications which may alter heart rate, blood pressure or cardiac output
21. Previous history of middle ear equalization problems at discretion of PI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Sequence matched median PaO2 per dose cohort comparing TSC vs PBO | Up to 10 ± 1 minutes after final VO2 max
  Comparison of partial pressure of oxygen (PaO2) at altitude between control and experimental exposures
Sequence matched median VO2 per dose cohort comparing TSC vs PBO | Up to 33 minutes (achievement of peak wattage)
  Comparison of maximal oxygen consumption (VO2 max) at altitude between control and experimental exposures

SECONDARY OUTCOMES:
Effect of TSC on Median Oxygen Saturation | Up to 33 minutes (achievement of peak wattage)
  Comparison of oxygen saturation (SpO2) between the control and experimental exposures
Effect of TSC on Median Serum Lactate Concentration | Up to 33 minutes (achievement of peak wattage)
  Comparison of lactate between the control and experimental exposures

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No